CLINICAL TRIAL: NCT03157609
Title: Paediatric Thermometry: Can the SpotOn™ Zero-Heat-Flux-Thermometry Sensor Accurately Measure Core Temperature in Children?
Brief Title: Can the SpotOn™ Zero-Heat-Flux-Thermometry Sensor Accurately Measure Core Temperature in Children?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SpotOn v 1.0
Record Dates: First submitted 2017-04-19; First posted 2017-05-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2017-10

CONDITIONS: Hypothermia; Anesthesia; Hypothermia Following Anesthesia; Children
Keywords: Thermometry; SpotOn
MeSH Terms: conditions — Hypothermia | interventions — Thermometry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: use of a third person (blinded to study design, population and statistics) which will extract data blindly from the hospital anaesthesia electronic database
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thermometry with SpotOn (Experimental): Application of SpotOn sensor on forehead.
  Interventions: Device: Thermometry
- Thermometry with oesophageal probe (Active Comparator): Nasal insertion of oesophageal temperature probe in the lower fourth of the oesophagus.
  Interventions: Device: Thermometry

INTERVENTIONS:
Device: Thermometry — Within the same patient comparison of 2 thermometry methods: SpotOn skin sensor versus oesophageal temperature probe

SUMMARY:
The present study aims to assess the accuracy of the SpotOn™ Zero-heat-flux-thermometry sensor in measuring core temperature in the paediatric population in the perioperative period.

DETAILED DESCRIPTION:
Temperature regulation in the perioperative period is of primordial importance in paediatric population - a particularly sensitive group for thermal variations.

In fact, infants lose a significantly high percentage of their core heat from skin perspiration in comparison to adults (where it approximates roughly 10%). This percentage can go up to 20% in premature infants and relates to the fact that cutaneous heat loss is "grosso modo" proportional to body surface area.

This higher thermal vulnerability is aggravated during the perioperative period, where body exposure to the cold operating room environment is increased, and where anaesthetic interventions impair the compensatory mechanisms to the extent of being unable to sufficiently increase heat production to compensate for hypothermia.

An alternative thermometry method called Zero-heat-flux was developed in the 1970's in an attempt to compensate for the limitations of pure skin temperature, while maintaining its practical character. It is based on the principle that the temperature 1-2 cm below skin surface reasonably approximates core temperature. In order to measure it, it uses 4-layered probe, with the following inside-out structure: patient temperature thermistor, insulating foam layer, heating (flex) circuit, and insulating foam. A servo-controlled system actively warms the probe circuit to the point where, theoretically, temperature equilibrium is achieved between the skin and deeper structures and there is zero heat transfer to the surrounding areas. This concept is commonly exemplified as the creation of a vertical isothermal tunnel between the skin surface and lower dermal layers. Assuming a good tissue perfusion, dermal temperature will reasonably approximate core temperature.

Although a systematic adult population validation is on its way, no data on the paediatric patients exists.

Considering the practical and non-invasive character of this skin surface probe, as well as the abovementioned thermal sensitivity concerns on the paediatric population, it seems that, should the probe indeed prove to be accurate in this age range, it can definitely contribute to the improvement of the perioperative temperature management in children.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II
* Age: 1d - 16 years
* Elective surgery
* Minimum anaesthesia time of 30 minutes

Exclusion Criteria:

* Fragile skin state in the forehead
* Know allergy to probe adhesive
* Maxillofacial trauma or lesions
* Procedures impeding proper use of SpotOn™ sensor (mostly maxillo-facial)
* Abnormal oesophageal anatomy/gastroesophageal procedures.
* Coagulopathy
* Neurologically impaired children with abnormal thermoregulation
* Extensive Haemodynamic instability
* Need for Vasopression
* Procedures associated with extended use of rinsing fluids (abdominal/thoracic lavages)
* Thoracoscopic/thoracotomic procedures (oesophageal probe cooling)
* Need for use of "over body" forced air warming systems
* Malignant Hyperthermia or family history of malignant hyperthermia
* Fever / Infectious patient
* All conditions that might be judged to alter skin perfusion in an abnormal way
* Anatomical variants (overt hydrocephalus …)
* Calibration/device failure

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Determination of accuracy of SpotOn in children | 2 hours
  degrees centigrade

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Carvalho, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Nadia Najafi, MD, Study Chair — Universitair Ziekenhuis Brussel; Jan Poelaert, PhDMD, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No